CLINICAL TRIAL: NCT01431105
Title: Phase I/IIa Study of Pharmacokinetics and Safety of Atorvastatin in Children With Coronary Artery Abnormalities Secondary to Kawasaki Disease
Brief Title: Pharmacokinetics (PK)/Safety Study of Atorvastatin in Children With Kawasaki Disease and Coronary Artery Abnormalities
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Children's Hospital Colorado (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Jane C. Burns MD, Chief, Division of Allergy, Immunology, Rheumatology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD-Atorvastatin
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atorvasatin (Experimental): Atorvastatin dose titration to maximum tolerated dose
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin dose titration to maximum tolerated dose (once daily for 6 weeks)
  Other Names: Lipitor

SUMMARY:
Kawasaki disease (KD) is the leading cause of acquired heart disease in children in the developed world. Despite available treatment, 25% of children in San Diego County appropriately treated for KD develop coronary artery abnormalities that could lead to complications later in life, including heart attack. Although investigators can identify children with KD that have these coronary artery abnormalities, there is no approved additional treatment to decrease coronary artery inflammation and arrest or prevent damage to the coronary arteries. Inflammation and damage to the arterial wall is central to these coronary artery abnormalities. Statins, a class of drugs that is known for lowering cholesterol, have also been shown to decrease inflammation in general as well as at the level of the vessel wall. Therefore, the investigators propose to study the safety of the drug atorvastatin in children with coronary artery abnormalities from KD.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 2 years to 17 years old
2. Meets clinical criteria for KD according to American Heart Association guidelines (Table 2): Fever (T≥38oC or 100.4oC) ≥ 3 days and ≥ 2 clinical criteria with left anterior descending coronary artery/right coronary artery z-score ≥ 2.5 or an aneurysm (≥ 1.5 x the adjacent segment) of one of the coronary arteries
3. Patient presents within the first 20 days after fever onset
4. Parent or legal guardian able and willing to provide informed consent and subject willing and able to provide assent when appropriate.
5. Post-menarchal females: Negative pregnancy test at screening and willing to use two forms of contraception during the study
6. Males engaging in sexual activity that could lead to pregnancy must use a condom.

Exclusion Criteria:

1. Use of a statin, fibrate, or niacin within the 3 months prior to enrollment
2. Have any chronic disease, except asthma, atopic dermatitis, autism or controlled seizure disorder
3. Screening creatine phosphokinase (CK) ≥ 3x upper limit of normal for age
4. Patient taking a CYP3A4 inhibitor (ie. cyclosporine or clarithromycin) in the last 7 days
5. Patient has a history of allergy to atorvastatin or its derivatives

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Burns, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Derived] He M, Chen Z, Martin M, Zhang J, Sangwung P, Woo B, Tremoulet AH, Shimizu C, Jain MK, Burns JC, Shyy JY. miR-483 Targeting of CTGF Suppresses Endothelial-to-Mesenchymal Transition: Therapeutic Implications in Kawasaki Disease. Circ Res. 2017 Jan 20;120(2):354-365. doi: 10.1161/CIRCRESAHA.116.310233. Epub 2016 Dec 6. PMID 27923814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atorvasatin
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atorvasatin
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 8
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34
Age [Median (Inter-Quartile Range); unit: years] — in years
  years | 4 [2.6 to 6.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SAE
Description: Number of participants who experienced an SAE within the 6 week study period
Time Frame: At 6 weeks after initiation of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Atorvasatin: Atorvastatin treated patients
Arm/Group | Atorvasatin
Number analyzed (Participants) | 34
Participants | 4

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Clinicaltrials.gov definition used for AEs
Arm/Group | Atorvasatin
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 4/34
Other Adverse Events (participants affected / at risk) | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvasatin (N=34)
Recrudescent Fever (Immune system disorders) | 2 (2) — Fever recurred consistent with recurrence of Kawasaki disease; this SAE was not attributable to the study drug
Worsening coronary artery aneurysm (Cardiac disorders) | 2 (2) — The coronary artery aneurysms worsened due to KD. These SAEs were not attributable to the study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvasatin (N=34)
Viral exanthem (Skin and subcutaneous tissue disorders) | 12 (12)
Constipation or Diarrhea (Gastrointestinal disorders) | 5 (5)
Bruising (Blood and lymphatic system disorders) | 15 (15)
Fever (Immune system disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT01431105/Prot_SAP_000.pdf